CLINICAL TRIAL: NCT00603811
Title: A Multicenter, Double-blind, Randomized, Escalating Dose-ranging Study to Investigate the Safety and Immunogenicity of the VAX102 Influenza Vaccine in Healthy Adults
Brief Title: Phase I Safety and Immunogenicity Study of VAX102 [Flagellin.HuM2e] Influenza Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VaxInnate Corporation (Industry)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAX102-01; Gates grant 42462
Record Dates: First submitted 2008-01-04; First posted 2008-01-29 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Influenza Infection
Keywords: Influenza vaccines; M2e
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): VAX102, a recombinant fusion protein that links the influenza A virus M2e antigen to S. typhimurium flagellin, a TLR5 ligand.
  Interventions: Biological: VAX102 [Flagellin.HuM2e]
- 2 (Placebo Comparator): Vaccine buffer
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VAX102 [Flagellin.HuM2e] — dose ranging, 2 i.m. doses given 28 days apart
  Arms: 1
Biological: Placebo — Placebo
  Arms: 2

SUMMARY:
This study will evaluate the safety and immunogenicity of VAX102 [Flagellin.HuM2e], a recombinant, inactivated, subunit influenza vaccine given as a two dose regimen at a range of doses.

DETAILED DESCRIPTION:
VAX102 is a cross-protective influenza A vaccine based on a recombinant protein expressed in E. coli. The protein comprises Salmonella typhimurium flagellin type 2 (STF2; TLR5 ligand) fused to Human M2e. The active component of the VAX102 vaccine is manufactured by a standard fermentation process. Unlike the HA and NA viral proteins, the amino acid sequence of M2e has remained remarkably stable in all human influenza A virus isolates. Thus an influenza vaccine based on the M2e antigen could elicit cross-protective immunity against most human influenza A virus strains. VAX102 vaccine relies on a single cross-reactive influenza A virus antigen manufactured by a recombinant protein fermentation-production process.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-49 years inclusive who provide written informed consent to participate.
* Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits.

Exclusion Criteria:

* Presence of significant acute or chronic, uncontrolled medical or psychiatric illness
* Documented influenza infection in the 6 months prior to study entry.
* Presently receiving or history of receiving any medications or treatments that affects the immune system
* Acute disease within 72 hours prior to vaccinations Investigational product (test article) administrations will occur on Days 0 and 28 (± 3).
* In-clinic safety evaluations will be performed at screening, before each test article dose, and at Days 1, 7 (± 2), 14 (± 2), 29, 35 (± 2), 42 (± 2), 60 (± 2), 120 (± 7), and 180 (± 7).
* Completion of a Memory Aid for seven days following each vaccine dose will be requested of subjects for use in accurate recall of local and systemic reactions.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Safety (local and systemic reactogenicity, laboratory tests and AEs) | 6 months

SECONDARY OUTCOMES:
Immunogenicity after prime and boost (serum IgG to M2e antigen) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christine Turley, MD, Principal Investigator — UTMB
Locations (2):
- United States (2):
  - Johnson County Clinical Trials, Lenexa, Kansas
  - Sealy Vaccine Center, UTMB, Galveston, Texas